CLINICAL TRIAL: NCT05239494
Title: How Does DT1 Sphere Perform in Those Who Previously Dropped Out of Contact Lenses Due to Comfort or Dryness?
Brief Title: Dailies Total 1 Sphere Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Andrew Pucker, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-300008359
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Dry Eye; Contact Lens Complication
Keywords: Contact Lens; Dailies Total1; Dry Eye; Comfort
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: All participants will be assigned to wear Dailies Total 1 Sphere contact lenses. They will report to 3 in person visits over the course of one month.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Dailies Total1 (Experimental): All participants will be asked to wear Dailies Total1 for the duration of this study.
  Interventions: Device: DT1 Sphere Contact Lenses

INTERVENTIONS:
Device: DT1 Sphere Contact Lenses — Devices: Dailies Total 1 Sphere Contact Lenses

SUMMARY:
CL discomfort is a complex phenomenon that has been defined by the Tear Film and Ocular Surface Society in their seminal report on contact lens (CL) discomfort as a condition that results in "episodic or persistent adverse ocular sensation related to lens wear, either with or without visual disturbance resulting from reduced compatibility between the CL and the environment, which can lead to decreased wearing time and discontinuation of CL wear." A recent review by Pucker and Tichenor found that CL discomfort was the top reason for established CL wears to cease wearing CLs. This same review alarmingly found that the frequency of CL dropout was about 20% across the many studies aimed at evaluating this condition, which is surprising given the introduction of better soft CL materials and daily disposable CLs over the past 20 plus years.

Dailies Total1 (DT1), which is a relatively new daily disposable CL, is a commonly used trouble shooting CL for patients who have failed with other CLs because DT1 utilizes advanced material technology that is specifically aimed at improving CL comfort. While DT1 is commonly used in these struggling patients, the literature currently lacks a targeted study aimed at understanding the frequency of successfully refitting CL dropouts into this advanced CL. Thus, the purpose of this study is to determine the frequency that past CL wearers who failed because of dryness or CL discomfort who can comfortable wear DT1.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-40
* Past contact lens wearers who have best corrected 20/20 visual acuity or better
* Participants will have had to have worn contact lenses for at least 1 year in the past
* Dropped out of contact lenses in the past 2 years do to discomfort or dryness
* Scores of 3 or less on the SPEED questionnaire
* Be able to be refit into Dailies Total1 Sphere contact lenses
* Provide a glasses prescription that is less than 3-years-old

Exclusion Criteria:

* Past rigid contact lens wearers
* A past history of being diagnosed with dry eye or ocular allergies
* Known systemic health conditions that are known to alter tear film physiology
* History of viral eye disease
* History of ocular surgery
* History of severe ocular trauma
* History of corneal dystrophies or degeneration
* Having active ocular infection or inflammation
* Currently using isotretinoin-derivatives or ocular medication
* Pregnant or breast feeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Kannarr Eye Care, Pittsburg, Kansas
  - ProCare Vision Center, Granville, Ohio
  - The Southern College of Optometry, Memphis, Tennessee

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dailies Total1
Started | 60
Completed | 59
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dailies Total1
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 60
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 24 [18 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 59
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 51
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) Contact Lenses Comfort Scores
Description: The median visual analog scale (VAS) scores at the 1-month visit (-50 to +50 scale with scores greater than 0 being comfortable).
Time Frame: 1 month
Population: Subjects were recruited via clinic records, email and fliers, and they were pre-screened with an Institutional Review Board (IRB)- approved qualification questionnaire over the telephone. Adult, 18- to 40-year-old (inclusive), past CL wearers who had a Logarithm of the Minimum Angle of Resolution (logMAR) best-corrected visual acuity of 0.00 or better were recruited. Subjects were required to have worn CLs for at least 1year in the past.
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Dailies Total1
Number analyzed (Participants) | 60
Score on a scale | 44 [40 to 48]
Statistical Analysis 1: Comparison: Dailies Total1; This study used a ±50 VAS scale, with values in the positive and negative range indicating that the contact lenses were comfortable or uncomfortable, respectively. A score of zero on this scale indicated neutral CL comfort; Test type: Superiority; p < 0.001, Shapiro-Wilks; Median Difference (Final Values) = 0.001

2. Secondary Outcome: Likert Questionnaire
Description: Number of participants who were likely to refer the study contact lens to a friend.
Time Frame: One Month
Population: All subjects who completed the 1 month visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Dailies Total1
Number analyzed (Participants) | 60
Participants | 59

ADVERSE EVENTS:
Time Frame: Adverse events were observed over a 6 month time period.
Arm/Group | Dailies Total1
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT05239494/Prot_SAP_000.pdf